CLINICAL TRIAL: NCT02798250
Title: Safety of Overestimation of a Meal Insulin Bolus in the Context of Dual-hormone Closed-loop Operation - Part 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, M.D., Ph.D., Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CLASS-Safety study - Part 2
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Artificial pancreas; Closed-loop system; Postprandial glucose control; Hypoglycemia; Insulin; Glucagon
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Insulin Resistance | interventions — Insulin; Glucagon

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dual-hormone CL with overestimation of meal size category (Active Comparator): A regular size standardized meal of 45g of carbohydrates will be provided to the patient and the meal size will be overestimated by one category, which will result in a meal insulin bolus for a meal of 65g of carbohydrates.
  Interventions: Other: Dual-hormone closed-loop; Drug: Insulin; Drug: Glucagon; Device: Dexcom G4 Platinum glucose sensor; Device: Accu Chek Combo insulin pump
- Dual-hormone CL with adequate estimation of meal size category (Active Comparator): A regular size standardized meal of 45g of carbohydrates will be provided to the patient and the meal size will be adequately estimated, which will result in a meal insulin bolus for a meal of 35g of carbohydrates.
  Interventions: Other: Dual-hormone closed-loop; Drug: Insulin; Drug: Glucagon; Device: Dexcom G4 Platinum glucose sensor; Device: Accu Chek Combo insulin pump

INTERVENTIONS:
Other: Dual-hormone closed-loop — Interventions will be undertaken 1 to 5 days after sensor insertion. Subjects will be admitted at the research center at 7:00. Subject's pump will be substituted with the study pump and an additional pump containing glucagon will be installed. At 7:00, closed-loop will be initiated. At 9:00, a standardized breakfast (45g CHO) will be served. Study subjects will consume the same meal on the two intervention days. During the intervention, patients will be allowed to do sedentary activities. Patients will be allowed to consume caffeine during the intervention, but will have to replicate their caffeine consumption on both interventions. The intervention day will end at 13:00.
Drug: Insulin — Participant's usual fast-acting insulin analog will be used: Lispro (Humalog), Aspart (NovoRapid) or Glulisine (Apidra).
Drug: Glucagon — Glucagon (Eli Lilly) will be used during dual-hormone closed-loop strategy.
Device: Dexcom G4 Platinum glucose sensor
Device: Accu Chek Combo insulin pump

SUMMARY:
In previous studies, investigators have studied if a pre-meal insulin bolus based on estimated carbohydrate meal size would alleviate the burden of carbohydrate counting without a significant degradation in postprandial glucose control. With this strategy, the patient would only have to evaluate the size of the meal in terms of carbohydrate (snack, regular, large or very large). It is however important to establish the safety of this simplified meal bolus approach. The safety of overestimating a meal insulin bolus in the context of closed-loop strategy needs to be assessed. For ethical reasons, only dual-hormone closed-loop will be tested.

Investigators hypothesize that dual-hormone closed-loop with overestimated meal size bolus will not increase time below 4.0 mmol/L compared to dual-hormone closed-loop with an adequately estimated meal size bolus.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years old.
2. Clinical diagnosis of type 1 diabetes for at least one year.
3. The subject will have been on insulin pump therapy for at least 3 months and currently using a fast acting insulin analog (Lispro, Aspart or Glulisine).
4. Last (less than 3 months) HbA1c ≤ 10%.
5. Currently using carbohydrate counting as the meal insulin dose strategy.

Exclusion Criteria:

1. Clinically significant microvascular complications: nephropathy (estimated glomerular filtration rate below 40 ml/min), neuropathy (especially diagnosed gastroparesis) or severe proliferative retinopathy as judged by the investigator.
2. Recent (< 3 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
3. Pregnancy.
4. Severe hypoglycemic episode within 1 month of screening.
5. Agents affecting gastric emptying (Motilium®, Prandase®, Victoza®, Byetta® and Symlin®) as well as oral anti-diabetic agents (Metformin, SGLT-2 inhibitors and DPP-4 inhibitors) if not at a stable dose for 3 months. Otherwise, these medications are acceptable and will be kept stable during the entire protocol.
6. Oral steroids unless patients present a low stable dose (e.g. 10 mg or less of prednisone per day or physiological doses, less than 35 mg/day, of hydrocortisone Cortef®). Inhale steroids at stable dose in the last month are acceptable.
7. Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator (e.g. unstable psychiatric condition).
8. Failure to comply with team's recommendations (e.g. not willing to change pump parameters, follow algorithm's suggestions, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-06; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Percentage of time below 4.0 mmol/L | The outcome measure will be calculated over the 4 hours following the breakfast meal. The 4-hour period is from 9:00 to 13:00.

SECONDARY OUTCOMES:
Mean glucose | The outcome measure will be calculated over the 4 hours following the breakfast meal. The 4-hour period is from 9:00 to 13:00.
Percentage of time of glucose concentrations between 4.0 and 8.0 mmol/L | The outcome measure will be calculated over the 4 hours following the breakfast meal. The 4-hour period is from 9:00 to 13:00.
Percentage of time of glucose concentrations between 4.0 and 10.0 mmol/L | The outcome measure will be calculated over the 4 hours following the breakfast meal. The 4-hour period is from 9:00 to 13:00.
Percentage of time of glucose concentrations below 3.1 mmol/L | The outcome measure will be calculated over the 4 hours following the breakfast meal. The 4-hour period is from 9:00 to 13:00.
Area under the curve of glucose values below 4.0 mmol/L | The outcome measure will be calculated over the 4 hours following the breakfast meal. The 4-hour period is from 9:00 to 13:00.
Area under the curve of glucose values below 3.1 mmol/L | The outcome measure will be calculated over the 4 hours following the breakfast meal. The 4-hour period is from 9:00 to 13:00.
Number of patients with at least one hypoglycemic event with or without symptoms | The outcome measure will be calculated over the 4 hours following the breakfast meal. The 4-hour period is from 9:00 to 13:00.
Total number of hypoglycemic event below 3.1 mmol/L | The outcome measure will be calculated over the 4 hours following the breakfast meal. The 4-hour period is from 9:00 to 13:00.
Total carbohydrate intake for hypoglycemia correction | The outcome measure will be calculated over the 4 hours following the breakfast meal. The 4-hour period is from 9:00 to 13:00.
Total insulin delivery | The outcome measure will be calculated over the 4 hours following the breakfast meal. The 4-hour period is from 9:00 to 13:00.
Total glucagon delivery | The outcome measure will be calculated over the 4 hours following the breakfast meal. The 4-hour period is from 9:00 to 13:00.

CONTACTS AND LOCATIONS:
Overall Officials: Remi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada